CLINICAL TRIAL: NCT04043026
Title: Stratifying Clinical Risk in Patients With Atrial Fibrillation and Chronic Kidney Disease by Studying How Abnormalities in Clot Structure/Function and Lipoproteins Contribute to Thrombosis and Bleeding
Brief Title: The Effects of Renal Function and Atrial Fibrillation on Lipoproteins and Clot Structure/Function
Acronym: RALiC
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment due to COVID19 pandemic
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool Centre for Cardiovascular Science (Unknown); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Liverpool John Moores University (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, Wern Yew Ding, Clinical Research Fellow, University of Liverpool
Other Study IDs: UoL001456 - 4843
Record Dates: First submitted 2019-07-26; First posted 2019-08-02 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation; Chronic Kidney Disease
Keywords: Anticoagulation; Fibrin clot structure and function; Lipids; Lipoproteins; Statin
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency, Chronic | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- WP1: AF + CKD: Anticoagulated participants with atrial fibrillation and chronic kidney disease
- WP1: AF + no CKD: Anticoagulated participants with atrial fibrillation and no chronic kidney disease
- WP1: no AF + CKD: Anticoagulated participants with chronic kidney disease and no atrial fibrillation
- WP1: no AF + no CKD: Anticoagulated participants without atrial fibrillation or chronic kidney disease
- WP2: AF + CKD: Anticoagulated participants with atrial fibrillation and chronic kidney disease, and are commencing statin therapy
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Statin — Any statin therapy
  Groups: WP2: AF + CKD

SUMMARY:
This study is designed to investigate the role of lipids/lipoproteins as a potential cause for the harmful changes seen in fibrin clot properties with renal dysfunction and atrial fibrillation

DETAILED DESCRIPTION:
This is a prospective, observational, blinded study that will be conducted in two parts. The first study will assess the relationship between lipids/lipoproteins and fibrin clot properties among anticoagulated atrial fibrillation patients with and without renal dysfunction. The second study will assess the effects of statin therapy on lipids/lipoproteins and fibrin clot properties in anticoagulated atrial fibrillation patients with renal dysfunction. Renal dysfunction is defined as an estimated glomerular filtration rate below 50 ml/min/1.73m2 for the purposes for this trial.

ELIGIBILITY:
6.1 Inclusion criteria

WP1:

* On anticoagulation therapy
* Informed consent obtained

WP2:

* Not receiving statins prior to recruitment
* Diagnosed atrial fibrillation
* On anticoagulation therapy
* Estimated glomerular filtration rate of <50 ml/min/1.73m2
* Informed consent obtained

6.2 Exclusion criteria

* Age <18 years
* Severe mitral stenosis or presence of metallic prosthetic valve
* Active or recent malignancy (<6 months)
* Active immunological disease
* Connective tissue disease
* Chronic liver disease
* Recent or chronic serious infection
* Chronic inflammatory disease
* Known haemophilia or thrombophilia
* Active bleeding
* Untreated hypothyroidism or hyperthyroidism
* Recent surgery (<3 months)
* Familial lipid disorders
* Concurrent use of steroids
* Dietary supplements known to influence lipids
* Contraindications/inability/unwillingness to commence statin (WP2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the hospital and specialist clinics in the community
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
WP1: Fibrin clot structure and function assessment using validated turbidity and fibrinolysis test | At baseline
  Lag time, maximum absorbance, time to maximum absorbance and clot lysis time
WP1: Fibrin permeation analysis using validated test | At baseline
  Permeation constant (Ks)
WP1: Low density lipoprotein fractions | At baseline
  Measure of low density lipoprotein subclass fractions
WP1: Oxidised low density lipoprotein | At baseline
  Measure of oxidised low density lipoprotein
WP2: Fibrin clot structure and function assessment using validated turbidity and fibrinolysis test | At baseline and after 6 weeks of statin therapy
  Lag time, maximum absorbance, time to maximum absorbance and clot lysis time
WP2: Fibrin permeation analysis using validated test | At baseline and after 6 weeks of statin
  Permeation constant (Ks)
WP2: Low density lipoprotein fractions | At baseline and after 6 weeks of statin
  Measure of low density lipoprotein subclass fractions
WP2: Oxidised low density lipoprotein | At baseline and after 6 weeks of statin
  Measure of oxidised low density lipoprotein

SECONDARY OUTCOMES:
WP1: Scanning electron microscopy | At baseline
  Qualitative assessment of fibril indices

CONTACTS AND LOCATIONS:
Overall Officials: Wern Yew Ding, Principal Investigator — University of Liverpool
Locations (2):
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: No